CLINICAL TRIAL: NCT07269418
Title: 160 / 5 000 Evaluation of the Result of Conoid Ligament Reconstruction According to an Anatomical Index in the Arthroscopic Treatment of Acromioclavicular Disjunctions
Brief Title: Optimization of Conoid Anatomical Reconstruction During Ligamentoplasty for Acromioclavicular Disjunction
Acronym: ORACLE
Status: Active, not recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2019-06-035-P-GUINAND; ID-RCB 2023-A02062-43 (Other: ANSM)
Record Dates: First submitted 2025-09-22; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Acromioclavicular; Dislocation; Ligament Repair or Reconstruction
Keywords: anatomic ligament reconstruction; acromioclavicular disjunction
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, longitudinal, multicenter, observational cohort study conducted on a population of patients who underwent ligamentoplasty for an acromioclavicular dislocation and who agreed to be followed for a period of two years starting from the day of hospital discharge.

DETAILED DESCRIPTION:
The objective of this study is purely observational. This study modifies the normal doctor-patient relationship due to the need for additional evaluations aimed at assessing the long-term functional outcome of the intervention through the administration of questionnaires.

The study will be carried out in five centers : the Clinique de l'Union in Toulouse (Saint-Jean), the Niçois Institute of Sport and Arthrosis in Nice, the Confluent Private Hospital in Nantes, the Clinique du Cap d'Or in La Seyne-sur-Mer and the Savoie Metropole Hospital Center in Chambéry.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 60
* Patient who has been informed of the objectives and conditions of the study and who has not objected to participation
* Patient who has undergone reconstruction for an acute Rockwood stage 4 or 5 acromioclavicular dislocation and for whom elbow immobilization was required for 6 weeks (self-rehabilitation in the supine position is possible from day 15, without pendulum or adduction movements).

Exclusion Criteria:

* Time between trauma and ACL reconstruction greater than 10 days
* History of surgery or trauma to the operated shoulder
* History of acromioclavicular surgery or trauma to the contralateral shoulder
* History of shoulder stiffness
* Patient playing a contact sport (rugby, American football)
* Presence of severe acromioclavicular osteoarthritis
* Mental impairment or any other reason that may hinder understanding or strict application of the protocol
* Patient under legal protection, guardianship, or curatorship
* Patient already included in an interventional therapeutic trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient operated on for anatomic ligament reconstruction for an acromioclavicular disjunction
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Acromioclavicular reduction | Month 3
  The parameters measured and compared with the contralateral side will be :
  * The CC (coracoclavicular) distance measured on the anteroposterior Zanca view
  * The AC-DC distance(Acromial center line to dorsal clavicle)
  * The GC-PC distance (Glenoid center line to posterior clavicle) Assessment of the result of the intervention on the acromioclavicular radiological reduction 3 months post-operatively according to the quantitative radiographic parameters described by Zumstein.
  The reduction will be considered as:
  * Complete if the AC-DC and GC-PC distances on the operated side are equal to those on the healthy side, with a margin of less than 10%.
  * Partial if the AC-DC and GC-PC distances on the operated side are equal to those on the healthy side, with a margin between 10% and 20%.
  * Poor if the AC-DC and GC-PC distances on the operated side are equal to those on the healthy side, with a margin greater than 20%.

SECONDARY OUTCOMES:
Pain assessement | Month 24
  Progression of pain with the Self-Constant score.
  Self-Constant score explores several domains such as pain, activity, strength, and mobility(functional evaluation) :
  * Pain is assessed using a numerical scale ranging from 0 (no pain) to 10 (unbearable pain)
  * Professional and leisure activities are evaluated by the patient using a numerical scale ranging from 0 (no activities possible) to 10 (all activities possible)
  * Mobility: the ranges to be considered are those that are possible actively and without pain. Active anterior elevation, active abduction, and active external rotation are evaluated by the patient with reference to photographs showing the different levels of range of motion
  * Muscle strength is evaluated according to the patient's ability to lift a certain number of common objects (from a 500 g can to a 9 kg pack of water) The total score ranges from 0 to 100 points, with 100 indicating a normal shoulder and 0 indicating a completely deficient shoulder
Shoulder functional assessment with the the ACJI Score (Acromioclavicular Joint Instability Score) | Month 3
  Describe, over the 2 years following surgery, changes in shoulder function scores:
  The ACJI Score (Acromioclavicular Joint Instability Score) assesses acromioclavicular joint instability across five dimensions:
  * Spontaneous pain and pain on palpation (out of 20 points)
  * Activities of daily living (out of 10 points)
  * Aesthetics (out of 10 points)
  * Function (out of 25 points), including evaluation of range of motion (flexion, abduction, external rotation, internal rotation) and abduction strength at 90° abduction
  * Radiological findings (out of 35 points): post-traumatic osteoarthritis, vertical stability, and horizontal stability The final score ranges from 0 to 100, with 0 corresponding to almost no function and 100 to normal function.
Return to work | Month 24
  Time to return to work after discharge from hospital
Resumption of physical and sporting activities (with the Self-Constant score) | Month 24
  Describe, over the 2 years following the intervention, the time and level of resumption of physical and sporting activities with Self-Constant score ranges from 0 (deficient shoulder) to 100 (normal shouder).
  Self-Constant score explores several domains such as pain, activity, strength, and mobility (functional evaluation):
  * Pain is assessed using a numerical scale ranging from 0 (no pain) to 10 (unbearable pain)
  * Professional and leisure activities are evaluated by the patient using a numerical scale ranging from 0 (no activities possible) to 10 (all activities possible)
  * Mobility: the ranges to be considered are those that are possible actively and without pain. Active anterior elevation, active abduction, and active external rotation are evaluated by the patient with reference to photographs showing the different levels of range of motion
  * Muscle strength is evaluated according to the patient's ability to lift a certain number of common objects (from 500g can to 9kg pack of water)
Patient satisfaction | Month 24
  Overall Assessment of Patient Satisfaction : Patient satisfaction with their care and outcomes will be assessed at the end of the study on a simple numerical scale ranging from 0 (very dissatisfied) to 10 (very satisfied).
Shoulder Functional assessment with the SSV Score (Subjective Shoulder Value Score) | Month 24
  Describe, over the 2 years following surgery, changes in shoulder function scores : The SSV Score (Subjective Shoulder Value Score) is a subjective assessment score that allows the patient to evaluate the value of their affected shoulder compared to a completely healthy shoulder. The result is expressed as a percentage (between 0 % and 100%, 0 is an anormal function and 100% a normal function of the shoulder).
Resumption of physical and sporting activities with the ACJI score | Month 3
  Describe, over the 2 years following the intervention, the time and level of resumption of physical and sporting activities with the ACJI score (acromioclavicular joint instability score).
  The ACJI Score (Acromioclavicular Joint Instability Score) assesses acromioclavicular joint instability across five dimensions:
  * Spontaneous pain and pain on palpation (out of 20 points)
  * Activities of daily living (out of 10 points)
  * Aesthetics (out of 10 points)
  * Function (out of 25 points), including evaluation of range of motion (flexion, abduction, external rotation, internal rotation) and abduction strength at 90° abduction
  * Radiological findings (out of 35 points): post-traumatic osteoarthritis, vertical stability, and horizontal stability The final score ranges from 0 to 100, with 0 corresponding to almost no function and 100 to normal function.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de l'Union, Saint-Jean, France